CLINICAL TRIAL: NCT04029545
Title: A Multicenter, Double-blind, Randomized, Controlled, Roll-over Retreatment Study of the Safety and Pain Associated With Injections of PN40082, RV001 With Topical Anesthetic or RV001 for Lip Augmentation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was placed on hold for the FDA review of revisions of the protocol. Review time resulted in roll-over subjects to be out of window for enrollment.
Sponsor: Prollenium Medical Technologies Inc. (Industry)
Collaborators: Symbio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO 2019-02
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-05

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Intervention Model Description: This is a multicenter, double-blind, randomized, controlled, roll-over retreatment clinical study of retreatment of subjects seeking lip augmentation who received treatment with either PN40082 or Restylane Silk in prior Protocol PRO 2018-02 (NCT04032977), and PN40082 in prior Protocol PRO 2018-03 (NCT04029519). Subjects meeting the inclusion/exclusion criteria will receive a single additional treatment with either RV001, RV001 with a topical anesthetic, or PN40082. The Evaluating Investigator will be blinded to the treatment. Injections of the study device will be performed by an unblinded Treating Investigator.
Who Masked: Participant, Outcomes Assessor
Masking Description: Injections of the study device are performed by the unblinded Treating Investigator. The blinded Evaluating Investigator is not allowed to retrieve study supplies or to be present during opening of the study supplies or during the injections. The Treating Investigator is not to have any discussion with the Evaluating Investigator or subjects regarding the treatments.
  Subjects are blinded to treatment assignment. Subjects are physically masked (blindfolded) just prior to and during all injection procedures to prevent observation of the syringes containing study device.
  Subjects, investigators, the Sponsor's staff conducting the study, and members of the administrative team will not have access to individual subjects' treatment assignments. In the event of an emergency that requires breaking of the study blind, the randomization code will be maintained by each investigator that can be opened to reveal the study device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- PN40082 (Experimental): PN40082 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w. The study device will be provided by the Sponsor.
  Interventions: Device: PN40082
- RV001 with lidocaine cream (Active Comparator): RV001 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid to be used with LMX4, a topical lidocaine. The study device will be provided by the Sponsor. LMX4 will be provided in commercial stock packaging by the Sponsor
  Interventions: Device: PN40082
- RV001 (Experimental): RV001 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid to be used alone. The study device will be provided by the Sponsor.
  Interventions: Device: PN40082

INTERVENTIONS:
Device: PN40082 — 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w.

SUMMARY:
The purpose of this study is to evaluate the safety of repeat injections and pain associated with injection of PN40082 and comparative pain associated with RV001 with a topical anesthetic and RV001 for lip augmentation.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, controlled, roll-over retreatment clinical study of retreatment of subjects seeking lip augmentation who received treatment with either PN40082 or Restylane Silk in prior Protocol PRO 2018-02 (NCT04032977), and PN40082 in prior Protocol PRO 2018-03 (NCT04029519). Subjects meeting the inclusion/exclusion criteria will receive a single additional treatment with either RV001, RV001 with a topical anesthetic, or PN40082. The Evaluating Investigator will be blinded to the treatment. Injections of the study device will be performed by an unblinded Treating Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Completed Protocol PRO 2018-03 OR Protocol PRO 2018-02 and did not enroll in Protocol PRO 2018-03.
2. Men or non-pregnant or non-breastfeeding women over 21 years of age
3. At PRO 2018-02 baseline visit had an overall score of very thin, or thin on the LFGS, as agreed upon by the Treating and Evaluating Investigators, and desires at least a 1-point improvement in overall LFGS score; OR Had a Fitzpatrick skin phototype IV, V or VI and has an LFGS score of thick or full, as agreed upon by the Treating and Evaluating Investigators, and desires treatment to the vermilion body of 1 or both lips
4. If female and of childbearing potential, a negative urine pregnancy test at Visit 1/Day 1 and the subject agrees to use adequate contraception during the study period.
5. Willing to give written informed consent.

Exclusion Criteria:

1. Women who are pregnant, lactating, or planning a pregnancy.
2. Subjects with a known history of allergy, anaphylaxis or hypersensitivity to injectable hyaluronic acid products, local anesthetics of the amide type such as lidocaine, or to latex.
3. Subjects with a significant ongoing adverse event from PRO 2018-02 or PRO 2018-03 that in the opinion of the investigator could be worsened by participation in this study.
4. Subjects that experienced an SAE, AESI, visual changes or other serious medical conditions during PRO 2018-02 or PRO 2018-03
5. Subjects who are unable to withhold thrombolytics, or inhibitors of platelet aggregation or nonsteroidal anti inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or gingko) within 10 days before AND after any injection session.
6. Subjects with clinically significant organic disease including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, preclude participation in the trial.
7. Subjects with lip tattoos, piercings, facial hair, or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments.
8. Subjects with abnormal lip function, with inability to effectively sip water through a straw.
9. Subjects with abnormal lip sensation with inability to feel a 0.4G monofilament or a cotton wisp at any site on the lip.
10. Subjects with moderate or severe abnormal lip asymmetry.
11. Subjects with any mass formation on the lip.
12. Subjects with dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities as judged by the Treating Investigator. Subjects planning to undergo extensive dental procedures such as dental implants, multiple tooth extractions, or oral surgery should not participate. Minor dental procedures such as teeth cleaning and repair of caries are not exclusionary.
13. Subjects that have undergone facial plastic surgery or received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene, polyacrylamide, lifting threads) anywhere in the face or neck, or are planning to be implanted with any of these products during the study.
14. Subjects that have undergone semi-permanent dermal filler treatment (e.g., calcium hydroxylapatite, poly-L-lactic acid) in the lower face (below the orbital rim) within 12 months before enrollment or are planning to undergo such treatment during the study.
15. Subjects that have undergone facial tissue augmentation with fat injections, botulinum toxin injections in the lower face (below the orbital rim), mesotherapy, or cosmetic procedures in the face or neck (e.g., face-lift, laser, photo-modulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, microneedling, or other ablative procedures) within 9 months before enrollment or are planning to undergo any of these procedures during the study.
16. that have used ANY lip filling agents within 12 months of study enrollment (hyaluronic acid products, collagen-based products, etc.) other than Investigational Device administered in PRO 2018-02 and PRO-2018-03.
17. Subjects that have used any lip plumping products or devices within 10 days before enrollment or are planning to use such products during the study.
18. Subjects that have begun using any over-the-counter (OTC) or prescription oral or topical anti wrinkle products for the lips or around the mouth within 90 days before enrollment or are planning to begin using such products during the study (Subjects who have been on a stable regimen of such products for at least 90 days are eligible for the study and must continue their regimen throughout the study).
19. Subjects that have a history or presence of bleeding disorders.
20. Subjects that have used systemic corticosteroids or immunosuppressive medications within 30 days prior to treatment.
21. Subjects that are on a concurrent regimen of lidocaine or structurally related local anesthetics (e.g., bupivacaine)
22. Subjects that have an active inflammation (skin eruptions such as cysts, pimples, rashes, or hives), infection cancerous or precancerous lesion, or unhealed wound on the face.
23. Subjects that have a history of known susceptibility to keloid formation or hypertrophic scars.
24. Subjects that have porphyria.
25. Subjects that have active herpes labialias lesions at the time of injections. Subjects with a history of herpes labialis who have had four (4) or more outbreaks in the 12 months prior to enrollment are also excluded even in the absence of lesions at the baseline visit.
26. Subjects that have impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction that, in the opinion of the investigator, would place them at risk of associated complications from these illnesses during the course of the study.
27. Subjects that have any uncontrolled disease, i.e., a condition that has not been appropriately diagnosed, evaluated, and received medically appropriate treatment or care
28. Subjects that have severe cardiovascular disease; examples include but are not limited to New York Heart Association heart failure classification III or IV, unstable angina, and internal pacemakers. Potential subjects with other significant cardiovascular diseases should be discussed with the Medical Monitor before enrolling.

    -

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy R Smith, MD, Study Director — California Dermatology & Clinical Research Institute
Locations (5):
- United States (5):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - International Dermatology Research, Inc, Miami, Florida
  - Skin Specialists, PC, Omaha, Nebraska
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Skintastic, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PN40082: PN40082 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w.
- RV001 With Lidocaine Cream: RV001 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid to be used with LMX4, a topical lidocaine.
- RV001: RV001 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid to be used alone.
Period: Overall Study
Arm/Group | PN40082 | RV001 With Lidocaine Cream | RV001
Started | 2 | 1 | 2
Completed | 2 | 1 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PN40082 | RV001 With Lidocaine Cream | RV001 | Total
Number analyzed (Participants) | 2 | 1 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 50.5 [40 to 61] | 55 [55 to 55] | 58 [52 to 64] | 54.4 [40 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 1 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved Pain Score From Baseline at Visit 2
Description: Compare subject pain scores with a 100 mm visual analog scale with 00 being no pain (better outcome) and 100 being worst possible pain (worse outcome)
Time Frame: Visit 1/Day 1 through Visit 2/Month 1, 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | PN40082 | RV001 With Lidocaine Cream | RV001
Number analyzed (Participants) | 2 | 1 | 2
Participants | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Each subject will be monitored for the occurrence of AEs, including serious adverse events (SAEs), starting immediately after treatment initiation. Each subject will be followed for safety monitoring until he/she is discharged from the study, an average of 2 months. Follow-up procedures related to pregnancy, AEs, or SAEs may continue beyond the end of the study, up to 6 months.)
Arm/Group | PN40082 | RV001 With Lidocaine Cream | RV001
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Five subjects were enrolled. The study was placed on hold for the revision of the protocol. After the revision was completed, all eligible subjects had missed the time frame for inclusion in the study. The 5 subjects completed the study. No statistical analysis was performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04029545/Prot_SAP_002.pdf